CLINICAL TRIAL: NCT02852434
Title: Self-administered Lidocaine Gel for Pain-control During Cervical Preparation for Dilation and Evacuation: A Randomized Controlled Trial
Brief Title: Self-administered Lidocaine Gel for Pain-control During Cervical Preparation for Dilation and Evacuation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-38200
Record Dates: First submitted 2016-06-20; First posted 2016-08-02 (Estimated); Results first posted 2018-04-17 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Pain Management, Cervical Preparation
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self-administered Gel (Experimental): Patient-administered, vaginal lidocaine gel (2%)--inserted 15 minutes prior to cervical preparation procedure
  Interventions: Drug: Lidocaine Gel (2%)
- Paracervical Block (Active Comparator): Provider-administered lidocaine (1%) paracervical injection--administered immediately prior to tenaculum placement
  Interventions: Drug: Lidocaine Paracervical Block (1%)

INTERVENTIONS:
Drug: Lidocaine Gel (2%)
  Arms: Self-administered Gel
Drug: Lidocaine Paracervical Block (1%)
  Arms: Paracervical Block

SUMMARY:
This study seeks to compare self-administered lidocaine gel for pain control during cervical preparation for dilation and evacuation (D&E) to paracervical block.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 and older
* Intrauterine pregnancy ≥16 weeks gestation
* English speaking competency
* Willing and able to sign consent forms
* Agree to comply with study procedures

Exclusion Criteria:

* Women less than 18 years of age
* IV conscious sedation
* Known allergy to study medication (lidocaine)
* Any women not meeting inclusion criteria above will be excluded from participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, MD, MS, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schivone GB, Lerma K, Montgomery C, Wright P, Conti JA, Blumenthal PD, Shaw KA. Self-administered lidocaine gel for local anesthesia prior to osmotic dilator placement: a randomized trial. Contraception. 2019 Mar;99(3):148-151. doi: 10.1016/j.contraception.2018.11.013. Epub 2018 Nov 27. PMID 30500336

RESULTS

PARTICIPANT FLOW:
Groups:
- Self-administered Gel: Patient-administered, vaginal lidocaine gel (2%)--inserted 15 minutes prior to cervical preparation procedure
  Lidocaine Gel (2%)
- Paracervical Block: Provider-administered lidocaine (1%) paracervical injection--administered immediately prior to tenaculum placement
  Lidocaine Paracervical Block (1%)
Period: Overall Study
Arm/Group | Self-administered Gel | Paracervical Block
Started | 36 | 36
Completed | 34 | 35
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Unsuccessful Dilator Procedure | 2 | 0

BASELINE CHARACTERISTICS:
Population: Participants who completed the protocol are included in the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Self-administered Gel | Paracervical Block | Total
Number analyzed (Participants) | 34 | 35 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.7 (7.87) | 27.2 (7.14) | 27.9 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 35 | 69
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 12 | 23
  Not Hispanic or Latino | 22 | 23 | 45
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 9 | 23
  White | 14 | 19 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 7 | 13
Region of Enrollment [Number; unit: participants]
  United States | 34 | 35 | 69
Gestational Age [Median (Full Range); unit: weeks] | 19 [16 to 23.4] | 19.4 [16 to 24] | 19.2 [16 to 24]

OUTCOME MEASURES:

1. Primary Outcome: Pain Perceived at the Time of Laminaria or Osmotic Dilator Insertion
Description: Measured by visual analogue scale (VAS), 0-100; Pain was measured on a 100 mm VAS scale. Lower scores correspond to less pain, higher scores correspond to more pain.
Time Frame: Intraoperative; Immediately (0-30 seconds) following cervical dilation
Population: Participants who completed the protocol are included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Self-administered Gel | Paracervical Block
Number analyzed (Participants) | 34 | 35
units on a scale | 48.4 (26) | 56.3 (29)

2. Secondary Outcome: Anticipated Pain Measured by Visual Analogue Scale
Description: Measured by visual analogue scale (VAS), 0-100, Pain was measured on a 100 mm VAS scale. Lower scores correspond to less pain, higher scores correspond to more pain.
Time Frame: Preoperative; 30 minutes prior to procedure
Population: Participants who completed the protocol are included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Self-administered Gel | Paracervical Block
Number analyzed (Participants) | 34 | 35
units on a scale | 47.2 (22) | 58.7 (18)

3. Secondary Outcome: Baseline Pain Measured by Visual Analogue Scale
Description: as for outcome 2
Time Frame: Immediately prior to procedure
Population: Participants who completed the protocol are included in the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Self-administered Gel | Paracervical Block
Number analyzed (Participants) | 34 | 35
units on a scale | 2.6 (55) | 6.6 (10)

4. Secondary Outcome: Speculum Placement Measured by Visual Analogue Scale
Description: as for outcome 1
Time Frame: Intraoperative; Immediately following speculum placement
Population: Participants who completed the protocol are included in the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Self-administered Gel | Paracervical Block
Number analyzed (Participants) | 34 | 35
units on a scale | 24.7 (22) | 31.2 (25)

5. Secondary Outcome: Overall Pain Measured by Visual Analogue Scale
Description: as for outcome 1
Time Frame: Postoperative; Assessed once 10 minutes after procedure
Population: Participants who completed the protocol are included in the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Self-administered Gel | Paracervical Block
Number analyzed (Participants) | 34 | 35
units on a scale
  Overall Pain | 45.4 (26.7) | 51.7 (25.7)
  Overall Experience | 65.2 (30) | 62.4 (30)
  Provider Reported Ease of Insertion | 27 (29) | 21 (22)

ADVERSE EVENTS:
Time Frame: 1 Day (day of procedure)
Description: No data were collected following the day of procedure; Participants who completed the protocol are included in the analysis.
Arm/Group | Self-administered Gel | Paracervical Block
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/35
Other Adverse Events (participants affected / at risk) | 0/34 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-18): https://cdn.clinicaltrials.gov/large-docs/34/NCT02852434/Prot_SAP_000.pdf